CLINICAL TRIAL: NCT04039646
Title: Enhanced Recovery After Surgery in Patients With Perforated Peptic Ulcer Disease Who Underwent Laparoscopic Repair, a Randomised Controlled Clinical Trial
Brief Title: ERAS in Patients With Perforated Peptic Ulcer Disease Who Underwent Laparoscopic Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Chairman of General Surgery, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RASS-01
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Hospital Stay; Hospital Cost
Keywords: Perforated peptic ulcer; Enhanced recovery after surgery; Laparoscopic repair; Complications
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard postoperative care group (Active Comparator): Patients received standard postoperative care as ususal.
  Interventions: Combination Product: ERAS treatment
- ERAS group (Experimental): Patients received postoperative ERAS treatment.
  Interventions: Combination Product: ERAS treatment

INTERVENTIONS:
Combination Product: ERAS treatment — The ERAS group had an enhanced postoperative recovery protocol. The gastric content was aspirated via the nasogastric tube by the anesthesiologist at the end of the procedure, and the nasogastric tube was withdrawn in the operating room immediately after the patient had recovered from anesthesia. and also early feeding and move.

SUMMARY:
Perforated peptic ulcer (PPU) is a frequent emergency condition worldwide with associated mortality up to 30%. Open procedures have in the most part been replaced by laparoscopic techniques. The standard postoperative management of PPUD patients is predominantly based on traditional practices. The aim of this randomized controlled clinical trial was to investigate the feasibility of enhanced postoperative recovery pathways in patients who underwent laparoscopic repair for Perforated peptic ulcer.

DETAILED DESCRIPTION:
Perforated peptic ulcer (PPU) is a frequent emergency condition worldwide with associated mortality up to 30%. Open procedures have in the most part been replaced by laparoscopic techniques. The standard postoperative management of PPUD patients is predominantly based on traditional practices. Randomization will be made at the end of the surgical procedure. Patients will be included in groups 1 or2. Group 1 is the control group and will receive standard postoperative care, and group 2 is the ERAS group.The aim of this randomized controlled clinical trial was to investigate the feasibility of ERAS in patients who underwent laparoscopic repair for Perforated peptic ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Perforated ulcer less than 10 mm in size
2. Patients received laprascopic repair

Exclusion Criteria:

-

1. refusal to join the study or sign the informed consent form 3. age younger than 18 years 3.the presence of any psychiatric or neurologic disease 4. class 3 and 4 surgical patients according to the classification of The American Society of Anesthesiologists 5. septic shock on admission 6. pregnancy 7. multiple perforated peptic ulcers 8. spontaneously sealed-off perforated ulcers that were diagnosed either preoperatively or during surgery and that did not require surgical repair 9.conversion to open technique 10. perforated ulcers that were not amenable to Graham patch repair because of size or technical considerations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Hospital stay | 30 days
  The time patients stay in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Li Hua Tian, Principal Investigator — Ethics center, Beijing Chaoyang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No